CLINICAL TRIAL: NCT06481423
Title: Digital Management of Sleep Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jia Xiu (Other)
Responsible Party: Sponsor-Investigator, Jia Xiu, Professor, Fudan University
Organization: Fudan University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FE22197I
Record Dates: First submitted 2024-06-20; First posted 2024-07-01 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Chronic Insomnia
Keywords: Digital cognitive behavior therapy for insomnia; Chronic Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Group (Experimental): Participants receive digital cognitive behavioral intervention for insomnia(dCBT-I) via their smartphone, and can freely access relaxing music in the app
  Interventions: Behavioral: dCBT-I; Behavioral: Relaxing music
- Control Group (Other): Participants can only freely access relaxing music in the app. They don't have access to dCBT-I
  Interventions: Behavioral: Relaxing music

INTERVENTIONS:
Behavioral: dCBT-I — A digital cognitive behavioral intervention course that addresses multiple aspects such as basic sleep knowledge, sleep hygiene, sleep behaviors, improving negative cognition, and improving emotions. The intervention is delivered through video, audio, and text formats.
  Arms: Intervention Group
Behavioral: Relaxing music — Participants can freely listen relaxing music

SUMMARY:
The goal of this clinical trial is to explore whether cognitive behavioral intervention for insomnia(CBT-I) realized through audio, video, and articles on smartphone apps("ForSleep" developed by the investigators) can improve the sleep quality of insomnia patients. The main question it aims to answer is:

Does CBT-I delivered via smartphone apps improve sleep quality evaluated by scales in patients with insomnia?

Investigators will compare the treatment group receiving the CBT-I intervention via smartphone apps to a control group receiving relaxation training to see if there are significant improvements in sleep quality.

Participants will be asked to:

Use an app("ForSleep") designed for CBT-I to follow a structured therapy program.

Complete daily sleep diaries and periodic scales to track their sleep quality.

DETAILED DESCRIPTION:
All participants sign the informed consent form online. The study is an online, single-blind, parallel-group, superiority randomized experiment of digital CBT-I(dCBT-I). The randomization is performed using stratified random sampling to ensure non-significant differences in age, gender, and basic sleep quality between the two groups. The screening, informed consent, assessments, allocation to conditions, delivery of the interventions, scale evaluations, and follow-ups are all carried out online. WeChat chatting groups for daily notification and communication are set up respectively. The experiment lasts 5 (and more) weeks included 3 weeks of intervention and 2 weeks of follow-up.

All participants are required to keep sleep diaries. They self-evaluate via Insomnia Severity Index (ISI), Dysfunctional Beliefs and Attitudes about Sleep (DBAS), Sleep Hygiene Index (SHI), and Epworth Sleepiness Scale (ESS) to assess insomnia severity, sleep-related cognition, and behaviors at 5 time points. The first 3 times are at the first day, after 7 days and 14 days, before starting each new session. After 3-week program, the above scales are retaken during days 22~25 and days 36~39 as follow-ups. The evaluating time is different on account of individual rate of progress to accomplish the 3-week program.

Digital cognitive behavioral therapy is delivered using an app developed by Fudan University. Digital intervention is structured into 3 sessions with a 7-days course in each session. The intervention group undertook 3 weeks of tasks which consisted of cognitive, behavioral, and relaxation parts of CBT-I and typically lasted 15 minutes per day. Two pieces of relaxing music are recommended daily to the control group instead of the standard relaxation practice. All participants have access to 30 relaxing music and articles on sleep hygiene that are made available in the app.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years old
* Insomnia Severity Index Scale (ISI) score of 8~21
* Proficient in the use of smartphones
* Chinese native speaker

Exclusion Criteria:

* Those with other combined sleep problems, such as apnoea syndrome, restless leg syndrome, etc.
* Women during pregnancy
* risky jobs that require high concentration, such as working at heights, long-distance driving, etc.
* previous or current diagnosis of severe neurological disorders such as epilepsy
* previous or current diagnosis of mental illness such as depression, bipolar disorder, schizophrenia, obsessive-compulsive disorder, etc.
* history of drug or alcohol abuse
* a significant negative risk of suicide
* serious physical illness (e.g., cardiovascular, hepatic, renal, etc.)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 358 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Pittsburgh Sleep Quality Index Scale(PSQI) | baseline(before the intervention); intervention stage(every week during 3-week intervention); follow-up stage(every week during 2-week follow-up)
  A scale that evaluates sleep quality, the scale scores range from 0 to 21, and lower scores mean a better outcome

SECONDARY OUTCOMES:
Dysfunctional Beliefs and Attitudes about Sleep Scale(DBAS) | baseline(before the intervention); intervention stage(every week during 3-week intervention); follow-up stage(every week during 2-week follow-up)
  A scale that evaluates the sleep attitude, the scale scores range from 0 to 64, and lower scores mean a better outcome
Sleep Hygiene Index Scale(SHI) | baseline(before the intervention); intervention stage(every week during 3-week intervention); follow-up stage(every week during 2-week follow-up)
  A scale that evaluates sleep hygiene, the scale scores range from 0 to 52, and lower scores mean a better outcome
The Insomnia Severity Index Scale(ISI) | baseline(before the intervention); intervention stage(every week during 3-week intervention); follow-up stage(every week during 2-week follow-up)
  A scale that evaluates the severity of insomnia, the scale scores range from 0 to 28, and lower scores mean a better outcome
Epworth Sleepiness Scale(ESS) | baseline(before the intervention); intervention stage(every week during 3-week intervention); follow-up stage(every week during 2-week follow-up)
  A scale that evaluates sleepiness, the scale scores range from 0 to 24, and lower scores mean a better outcome

CONTACTS AND LOCATIONS:
Overall Officials: Shouyan Wang, PhD, Study Chair — Fudan University
Locations (1):
- Institute of Science and Technology for Brain-Inspired Intelligence, Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No
Due to concerns regarding patient confidentiality and privacy, the investigators are unable to share the data from our study. The sensitive nature of the data includes personal health information that could potentially identify individual participants. Despite our best efforts to anonymize the data, the risk of re-identification remains. Additionally, the investigators are bound by ethical guidelines and institutional policies that require us to protect the privacy of our participants and maintain the confidentiality of their information. As such, the investigators must restrict access to the data to ensure compliance with these ethical and legal standards.